CLINICAL TRIAL: NCT05099328
Title: Recasting and Book Reading Under Ideal (Dose-controlled) and Typical (Dose-variable) Conditions: The Role of Fidelity and Adherence in Production and Comprehension Outcomes for Children With DLD
Brief Title: Recasting or Book Reading by Parents or Clinicians
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Amanda J. Owen Van Horne, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 307878; R01DC018276 (NIH)
Record Dates: First submitted 2021-10-05; First posted 2021-10-29 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Developmental Language Disorder and Language Impairment
Keywords: Recasting; Book Reading; Parent Coaching; Syntax Stories; Theoretical Domains Framework; Complex Syntax; Expressive language; Language Intervention
MeSH Terms: conditions — Language Development Disorders; Language Disorders

STUDY DESIGN:
Intervention Model Description: Children are stratified based on treatment site. Then they are randomly assigned to receive treatment for 1 of 2 targets, using 1 of 4 methods of intervention. Each child is randomly assigned to parent or clinician delivered intervention using books or recast therapy (2x2 design). Then assignment to treatment targets is assigned so that it is evenly distributed within each condition.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor is unaware of the arm to which the child has been assigned and is also unaware of which of two targets are the treatment target.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Recast Therapy Provided By Clinician (Experimental): Children will be exposed to recasts at a rate of 1/minute. Treatment will be provided 2x/week for 8 weeks for a total of 16 visits (960 recasts). 2 additional weeks are allocated for make up visits. Treatment will be provided by a trained, certified, licensed Speech Language Pathologist (SLP).
  Interventions: Behavioral: Recast Therapy
- Illustrated Syntax Stories Provided by Clinician (Experimental): Children will be listen to books that are specially scripted to promote the use of a particular syntax target. Treatment will be provided 2x/week for 8 weeks for a total of 16 visits (960 exposures), with 2 books read at each visit. 2 additional weeks are allocated for make up visits. Treatment will be provided by a trained, certified, licensed SLP.
  Interventions: Behavioral: Syntax Stories
- Recast Therapy Provided by a Caregiver (Experimental): Caregivers will receive two training sessions on how to provide recast therapy and demonstrate their skill at providing recast therapy with support from the clinician. Caregivers will then provide recast therapy at a rate of 1 recast per minute to their children for a minimum of 16 hrs (960 exposures) scheduled at their own convenience.
  Interventions: Behavioral: Recast Therapy
- Illustrated Syntax Stories Provided by a Caregiver (Experimental): Caregivers will receive two training sessions on how to provide read illustrated syntax stories to their children and demonstrate their skill at reading these stories with support from the clinician. Caregivers will then read these stories to their children for a minimum of 32 book readings (960 exposures)
  Interventions: Behavioral: Syntax Stories

INTERVENTIONS:
Behavioral: Recast Therapy — Recast therapy is when a interventionist uses the child's own productions as a platform for restating or recasting the child's speech with corrections or alterations to focus on a particular syntax target.
  Other Names: Focused Stimulation
  Arms: Recast Therapy Provided By Clinician; Recast Therapy Provided by a Caregiver
Behavioral: Syntax Stories — Syntax stories are specially constructed stories read verbatim designed to teach a syntax target.
  Other Names: Priming; Book Reading
  Arms: Illustrated Syntax Stories Provided by Clinician; Illustrated Syntax Stories Provided by a Caregiver

SUMMARY:
Developmental Language Disorder (DLD) affects approximately seven percent of the population and is characterized by grammatical deficits that cascade into lifelong academic challenges and under-employment. Current treatments for DLD produce good outcomes under ideal, high intensity conditions or when parents have been trained to deliver therapy using intense coaching methods; however, current publicly funded service delivery systems and private-pay reimbursement models do not support treatment being delivered in this ideal fashion for children older than three. This project will examine alternative methods of delivering treatment that may be more feasible under typical conditions and will identify implementation barriers, with the goal of improving long-term outcomes for children with DLD. We hypothesize that feasibility and palatability will influence dose, which will in turn affect the overall language outcomes.

ELIGIBILITY:
Inclusion Criteria:

Child with DLD

* Age: 4-9 years old
* Primarily English speaking: as documented by 20% or less exposure to another language, per parent report on the MAPLE
* Diagnosed with DLD as documented by standard score below 85 on the Diagnostic Evaluation of Language Variation - Norm Referenced (DELV-NR) composite, a dialect neutral assessment (Seymour, Roeper, de Villiers, & De Villiers, 2005).
* Nonverbal Intelligence Quotient (IQ) within typical range as documented by a t-score at or above 35 on the Developmental Abilities Scale (DAS), matrices similarities subscale, (Elliott, 2007).
* Hearing within the typical range: Pass screening at 25 dB for 1, 2, 4 kHz; OR scores within the typical range via SoundScouts hearing screening app; OR clear hearing assessment from an audiologist, otolaryngologist, medical doctor, or other professional.
* No diagnosis of Autism: Cutoff score of 15 on the Social Communication Questionnaire, (Rutter, Bailey, & Lord, 2003)
* No diagnosis of significant sensory-motor concerns or significant psychiatric disorders per parent report
* Able to benefit from treatment:

  * Score below 60% correct on experimenter developed elicited production probes of passives and object relative clauses
  * Producing simple transitive sentences (SVO) and mean length of utterance (MLU) of 2.5 on 100 utterance language sample

Caregiver

* Serves as the primary caregiver for an eligible child (may include grandparents, etc.)
* Basic literacy skills per self-report
* Willing to participate in caregiver training and caregiver-based treatments if child is assigned to that condition
* Willing to participate in questionnaires and structured interviews during post-test

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-08-28 (Estimated)

PRIMARY OUTCOMES:
Change in Accuracy on Elicited Production Probes | 2 week prior to the start of therapy; 2 week post therapy
  Children will respond to 20 item elicited production probes that ask the child to produce the treated structures and a control structure. Elicited Production Probes are highly reliable (ICC >.9), valid measures of children's use of a grammatical form. They have clinical relevance and align with the types of items that occur on standardized tests of language use.
Change in Comprehension probes (Proportion Looking) | 2 week prior to the start of therapy, 2 week post therapy
  Children will participate in an online looking while listening task with 24 items each for the treated target and a control (untreated) structure. Looks to areas of interest on the screen will be recorded. Proportion of time looking at the target picture will be the dependent variable. Looking patterns provide insight into the online processes associated with language comprehension and thus has the potential to inform future studies. These online measures have become well accepted as valid means of understanding comprehension. As far as we are aware there is limited psychometric data available for this age group, but Farris-Trimble & McMurray (2013) have shown these types of paradigms to be reliable.
Estimated Dose Delivered | During 10 week treatment period
  Adherence (attendance, reported therapy delivery)and treatment fidelity derived from recordings will be combined to estimate the number of exposures/recasts the caregiver provided to the child. This primary measure is important for future studies given the need to understand how well treatment is provided by parents and lab staff for these types of syntactic forms.
Semi-structured interviews | within 2 weeks post therapy ( ~12- 14 week mark in study timeline)
  Ethnographic interview examines the caregiver's comfort and understanding and motivation for participation in therapy. Ethnographic interviewing is a valid and reliable technique for qualitative data collection.

SECONDARY OUTCOMES:
Change in Comprehension probes (Pointing) | 2 week prior to the start of therapy, 2 week post therapy
  Children will participate in an online looking while listening task with 24 items each for the treated target and a control (untreated) structure. Points to the correct picture after the conclusion of eye gaze collection will be the dependent variable.
Palatability of treatment | During 10 week treatment period, immediately after each treatment session
  Likert ratings of how much therapy is enjoyed
Effortfulness of treatment | During 10 week treatment period, immediately after each treatment session
  Likert ratings of how effortful therapy is to deliver.
self-efficacy of treatment provider | During 10 week treatment period, immediately after each treatment session
  Likert ratings of how efficacious the provider perceived the activities to be
Caregiver grammar knowledge | In the first 1.5 weeks of the treatment period
  Written grammar quiz adapted from Brimo (in press). This questionnaire was previously validated for pre-service SLPs, early childhood educators, and practicing SLPs. The first two sections (implicit knowledge) have been used by Brimo. The last two sections (labeling) have been used in our lab to assess the knowledge of graduate clinicians.
Theoretical Domains Framework (TDF) Questionnaire | within 2 weeks post therapy ( ~12- 14 week mark in study timeline)
  Questionnaire aligned with Theoretical Domains Framework constructs that examines the caregiver's comfort and understanding and motivation for participation in therapy. This questionnaire was previously validated for providers of Physical Therapy.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Delaware, Newark, Delaware
  - University of Maryland, College Park, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Summary results of the primary outcomes for Aims 1 & 2 (elicited production and eye-gaze) will be uploaded within 12 months of the last data collection point for the final participant.
  We will track and provide information about participant flow. At each phase of participation, we will aggregate and report the following information:
  1. non-qualifiers: available screening information and reason for not continuing;
  2. qualifying participants who continue in the study: screening & pretest information, by treatment group;
  3. participants who complete the study: post-test scores, by treatment group;
  4. participants who drop out: reasons given for dropout, along with any adverse events;
  It is not possible to fully de-identify the interviews utilized in the mixed methods study (Aim 3). Thus, these data will not be shared. Additional data at the individual participant level may be sharable upon request and IRB approval for particular access.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 1 year after final data collection is complete
Access Criteria: IRB approval for access to data

DOCUMENTS (2):
  • Study Protocol (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT05099328/Prot_002.pdf
  • Informed Consent Form (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT05099328/ICF_003.pdf